CLINICAL TRIAL: NCT04641832
Title: The Effect of Chronic Cannabis Use on Neural Response to Acute Subconcussive Head Impacts
Brief Title: The Combined Effect of Chronic Cannabis Use and Subconcussive Head Impacts on Brain Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Keisuke Kawata, Assistant Professor, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2006187939
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Concussion, Mild
Keywords: soccer heading; subconcussive head impacts; cannabis
MeSH Terms: conditions — Brain Concussion; Marijuana Abuse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Dr. Kawata (PI) will only know subjects' group assignment and ensure blinded experiment and data processing. They will assign participants into two groups, chronic cannabis users and non-users. Group assignment will be based on self-reported cannabis use history and confirmed on 1st day of the study, with a saliva test ensuring no recent (24h-prior) use and a urine test to confirm history of chronic cannabis use or no use. Under the strict supervision of Dr. Kawata, experienced research assistants will perform soccer heading protocol, blood draws, neurocognitive and ocular-motor testing. Statistician will be blinded from group assignment. These processes will ensure single blind method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic cannabis use and subconcussive head impacts (Experimental): Group: Chronic cannabis users Criteria: self-reported chronic THC use (average use once per week but not dependent). Urine cannabis test must show positive.
  Device: Soccer Heading Soccer Heading: Subjects stood approximately 40 feet away from a JUGS soccer ball launcher and participated in 20 consecutive soccer headings, separated by one minute intervals.
  Interventions: Other: Soccer heading
- Non-cannabis use and subconcussive head impacts (Active Comparator): Group: Non cannabis users Criteria: self-reported none THC use. Urine cannabis test must show negative.
  Device: Soccer Heading Soccer Heading: Subjects stood approximately 40 feet away from a JUGS soccer ball launcher and participated in 20 consecutive soccer headings, separated by one minute intervals.
  Interventions: Other: Soccer heading

INTERVENTIONS:
Other: Soccer heading — A standardized and reliable soccer heading protocol will be used for the experiment. A triaxial accelerometer embedded in a head-band pocket and positioned directly below the external occipital protuberance (inion) to monitor linear and rotational head accelerations. A JUGS soccer machine will be used to simulate a soccer throw-in with a standardized ball speed of 25mph. The ball speed is similar to when soccer players make a long throw-in from the sideline to mid-field. Soccer players frequently perform this maneuver during practice and games. Subjects will stand approximately 40ft away from the machine to perform the heading. Participants perform 20 standing headers with 1 header per 30 seconds. The subjects will be instructed to direct the ball back toward the JUGS soccer machine in the air.

SUMMARY:
The purpose of this pilot study is to better understand the effects of chronic cannabis (THC) use on the neural responses to subconcussive head impacts, as a form of repetitive soccer headings. The study is designed to identify the physiological changes of cannabis using cohort (THC) and compare it to a nonusing cohort in order to see if the responses to 20 controlled bouts of soccer headings are exacerbated by the chronic cannabis use, diminished to less of a response, or unchanged, through an array of neurologic measures, including cognitive function, ocolar-motor function, autonomic function, and blood biomarkers. The hypothesis is that repetitive subconcussive head impacts will impair cognitive function in worse memory, attention span, and visual and verbal problem solving; this impairment will be greater in the chronic cannabis use groups than non-using group. The blood and salivary biomarkers neurofilament light (NFL) and glial fibrillary acidic protein (GFAP) will be measured in plasma, with the hypothesis that repetitive subconcussive head impacts will significantly increase plasma NFL and GFAP level at 24 hours-post heading and decrease by 72 hours-post heading, while remaining undetectable at 2 hours-post heading; the chronic cannabis use groups will see more severe effects on ocular-motor function than the non-using group. The study aims to determine the differences in acute effects of subconcussive head impacts on eye movement, attention, and language function between chronic cannabis use subjects and non-using subjects by evaluating ocular-motor function with near point of convergence and King-Devick tests. The hypothesis is that repetitive subconcussive head impacts will significantly increase impairments of eye movements, attention, and language function, as well as near point of convergence; the chronic cannabis use groups will see more severe effects on hampered ocular-motor function than the non-using group. Lastly, there is a cold pressor test to assess autonomic nerve function, with the hypothesis that repetitive subconcussive head impacts will decrease autonomic nerve function in chronic cannabis use patients to a greater degree than non-using subjects.

DETAILED DESCRIPTION:
NUMBER OF PEOPLE TAKING PART IN THE STUDY

We plan to recruit 45 THC using subjects and 45 non-using subjects.

PROCEDURES FOR THE STUDY

Participants will be assigned to the THC cannabis user group or the nonuser group based on participants' report of past cannabis use. These groups will then be verified using saliva and urine tests for cannabis use history.

The study consists of 4 test sessions during a 4-day period. The 1st day will take approximately 4 hours. The 2nd and 4th day will each take approximately 1 hour. Participants will not need to do anything on the 3rd day.

* The 1st test session takes place right before the soccer heading intervention.
* After the 1st test session, participants will then perform 20 soccer headings in 10 minutes.
* The 2nd test session takes place 2h after the intervention.
* The 3rd test session takes place approximately 24h after the intervention.
* The 4th test session takes place approximately 72h after the intervention.

During each test session, participants will be asked to complete a paper-pencil questionnaire assessing participants' current feeling. The questionnaire consists of 22 possible symptoms with 7-point scale to see if participants are experiencing concussion-related symptoms. A trained phlebotomist will draw blood from a vein in participants' arm at the four time points described in the above bulletpoints. Each 4mL blood sample is equivalent to approximately 1 teaspoon. A total of approximately 16mL (3-4 teaspoons) will be drawn during this study. The researchers will collect saliva samples (2mL) at each time point. Participants will be then asked to perform eye-movement tasks with directions from the research assistant. The eye-movement tasks consist of watching an object nearing the face (called a convergence test) and a brief test that asks participants to name numbers aloud from a screen. These eye-movement tasks will be repeated twice and will take about 2 minutes. After eye-movement testing, the investigators will ask participants to complete an imPACT test, which is a computerized test commonly used to diagnose concussions that measures memory, attention span, and visual and verbal problem solving. Completing the imPACT takes 20 to 25min. The last test is an autonomic function test, where participants will place participants' hand in a bowl of ice water for 60s while participants' heartrate is recorded.

The first 1st test session is slightly longer than the other two. It requires a saliva collection, where participants are asked to collect saliva in his/her mouth for approximately 15s before spitting onto a test strip. Researchers will need to collect about 7mL (1.5 teaspoon) of saliva from participants. This test will verify that participants have not used cannabis products in the past 72 hours. participants will also be asked for a urine sample. A urine sample of approximately 50mL will be used to verify cannabis use history over the past 3 months.

During the 1st day, after finishing the 1st test session, participants will perform 20 soccer headings. A standard size 5 soccer ball will be projected at 25 mph (equivalent speed to a long throw-in) by a JUGS soccer machine, and participants will perform 20 headers with 30 seconds resting period between each header. participants will be asked to direct the ball back towards the JUGS soccer machine in the air.

ELIGIBILITY:
Inclusion Criteria:

For Chronic THC User Group

1. being between 18 to 26 years of age
2. self-reported chronic THC use (average use once per week but not dependent)3) at least 3 years of soccer heading experience.

For Non-User Cohort

1. being between 18 to 26 years of age
2. self-reported non cannabis use in the past 6 months
3. at least 3 years of soccer heading experience

Exclusion Criteria:

1. any head, neck, or face injury in the 1 year prior to the study (e.g., concussion, eye injury);
2. history of vestibular, ocular, or vision dysfunction (e.g., macular degeneration)
3. currently taking any medications affecting balance (e.g., antibiotics)
4. pregnancy
5. HIV
6. any neurological disorders (e.g., seizure disorders, closed head injuries with loss of consciousness greater than 15 minutes, CNS neoplasm, spinal cord injury/surgery, history of stroke)
7. hypertension, cardiac arrhythmia, or pulmonary disease
8. lower extremity injury that would prohibit performing soccer headings
9. metal implants in the head

   Session-specific exclusion criteria will include:
10. used cannabis within the last 72 hours (verified by saliva cannabis test before intervention)
11. slept less than 4 hours before the 1st and 2nd test day (verified by screening questionnaire)
12. drank any alcoholic drinks or used recreational drugs 72 hours before the 1st test day and during the study period.
13. drank more than 3 cups of coffee before any test sessions
14. glasses are prohibited (contact lenses are okay) for safety purpose for the heading intervention

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Acute change in brain-derived blood and saliva biomarkers from pre to 24 hour post-heading | Blood samples will be collected at pre- and 24 hour post-heading
  Blood samples will be collected and centrifuged at 1500 x g for ten minutes at 4 degree celsius. Serum and saliva samples will be aliquoted and stored at -80 degree celsius until analysis.
  Serum and saliva samples will be assayed for S100B, neurofilament-light (NfL), glial fibrillary acidic protein (GFAP), and tau, and UCH-L1. All expression levels in pg/mL.
Acute change in brain-derived blood and saliva biomarkers from pre to 2 hour post-heading | Blood and saliva samples will be collected at pre- and 2 hour post-heading
  Blood samples will be collected and centrifuged at 1500 x g for ten minutes at 4 degree celsius. Serum and saliva samples will be aliquoted and stored at -80 degree celsius until analysis.
  Serum and saliva samples will be assayed for S100B, neurofilament-light (NfL), glial fibrillary acidic protein (GFAP), and tau, and UCH-L1. All expression levels in pg/mL.
Acute change in neurocognitive function from pre to 2 hour post-heading | Neurocognitive function will be assessed at pre- and 2 hour post-heading
  Participants will complete a computerized neurocognitive assessment (Immediate Post-Concussion Assessment and Cognitive Testing).
Acute change in neurocognitive function from pre to 24 hour post-heading | Neurocognitive function will be assessed at pre- and 24 hour post-heading
  Participants will complete a computerized neurocognitive assessment (Immediate Post-Concussion Assessment and Cognitive Testing).
Acute change in ocular-motor function from pre to 2 hour post-heading | Ocular-motor function will be assessed at pre- and 2 hour post-heading
  Participants will undergo 2 ocular-motor assessments: 1) near-point of convergence and 2) King-Devick Test--a brief assessment of saccadic eye movements, attention, and visual and language processing.
Acute change in ocular-motor function from pre to 24 hour post-heading | Ocular-motor function will be assessed at pre- and 24 hour post-heading
  Participants will undergo 2 ocular-motor assessments: 1) near-point of convergence and 2) King-Devick Test--a brief assessment of saccadic eye movements, attention, and visual and language processing.

SECONDARY OUTCOMES:
Acute change in brain-derived blood and saliva biomarkers from pre to 72 hour post-heading | Blood and saliva samples will be collected at pre- and 72 hour post-heading
  Blood samples will be collected and centrifuged at 1500 x g for ten minutes at 4 degree celsius. Serum and saliva samples will be aliquoted and stored at -80 degree celsius until analysis.
  Serum and saliva samples will be assayed for S100B, neurofilament-light (NfL), glial fibrillary acidic protein (GFAP), and tau, and UCH-L1. All expression levels in pg/mL.
Acute change in neurocognitive function from pre to 72 hour post-heading | Neurocognitive function will be assessed at pre- and 72 hour post-heading
  Participants will complete a computerized neurocognitive assessment (Immediate Post-Concussion Assessment and Cognitive Testing).
Acute change in ocular-motor function from pre to 72 hour post-heading | Ocular-motor function will be assessed at pre- and 72 hour post-heading
  Participants will undergo 2 ocular-motor assessments: 1) near-point of convergence and 2) King-Devick Test--a brief assessment of saccadic eye movements, attention, and visual and language processing.
Acute change in autonomic nerve function from pre to 2 hour post-heading | Autonomic response will be assessed at pre- and 2 hour post-heading
  Participants will undergo cold-pressor testing (CPT). CPT is a general assessment of the ability of the sympathetic nervous system to become activated. This test will be performed by submerging a participant's hand into cold water for 2 minutes while autonomic and hemodynamic variables are recorded. At each data collection, participants will be instrumented for the measurement of heart rate (electrocardiogram) and continuous blood pressure. Participants will rest quietly for ~10mins before the CPT begins. The test takes 2 minutes.
  Mean arterial pressure (in mm/Hg) is the outcome measure.
Acute change in autonomic nerve function from pre to 24 hour post-heading | Autonomic response will be assessed at pre- and 24 hour post-heading
  Participants will undergo cold-pressor testing (CPT). CPT is a general assessment of the ability of the sympathetic nervous system to become activated. This test will be performed by submerging a participant's hand into cold water for 2 minutes while autonomic and hemodynamic variables are recorded. At each data collection, participants will be instrumented for the measurement of heart rate (electrocardiogram) and continuous blood pressure. Participants will rest quietly for ~10mins before the CPT begins. The test takes 2 minutes.
  Mean arterial pressure (in mm/Hg) is the outcome measure.
Acute change in autonomic nerve function from pre to 72 hour post-heading | Autonomic response will be assessed at pre- and 72 hour post-heading
  Participants will undergo cold-pressor testing (CPT). CPT is a general assessment of the ability of the sympathetic nervous system to become activated. This test will be performed by submerging a participant's hand into cold water for 2 minutes while autonomic and hemodynamic variables are recorded. At each data collection, participants will be instrumented for the measurement of heart rate (electrocardiogram) and continuous blood pressure. Participants will rest quietly for ~10mins before the CPT begins. The test takes 2 minutes.
  Mean arterial pressure (in mm/Hg) is the outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Public Health, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
All study data will be included in publications.